CLINICAL TRIAL: NCT00286247
Title: Study to Determine the Efficacy and Safety of Docetaxel and Doxorubicin With INGN 201 in Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Introgen Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 201-010; MDACC ID-00-008
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Locally Advanced Breast Cancer (LABC)
MeSH Terms: interventions — advexin

INTERVENTIONS:
Genetic: INGN 201

SUMMARY:
A maximum of 60 subjects will be enrolled in the trial. It is a non-randomized, open label, single center study. All subjects undergo INGN 201 injection and IV chemotherapy: doxorubicin and docetaxel. This is done on the first 2 days of a 3-week cycle. After completion of 4 to 6 cycles, the subject either proceeds to surgery if the tumors respond to therapy, or goes off study if there is no tumor response.

ELIGIBILITY:
Documented late stage breast cancer: stage III A-B (excluding inflammatory breast carcinoma) or localized stage IV breast cancer

Male or female

18 years or older

Adequate bone marrow, liver, and kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States